CLINICAL TRIAL: NCT03383991
Title: Reverse Total Shoulder Arthroplasty Versus Hemiarthroplasty for Displaced 3- and 4-part Proximal Humeral Fractures in Patients Older Than 70 Years. A Multicenter Randomized Controlled Trial
Brief Title: Reverse Total Shoulder Arthroplasty Versus Hemiarthroplasty for Displaced 3- and 4-part Proximal Humeral Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Per Olerud, MD, PhD, Senior Consulting Orthopedic Surgeon, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 2013/1053-31/3
Record Dates: First submitted 2017-12-14; First posted 2017-12-27 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Humeral Fracture, Proximal
Keywords: Humeral Fracture, Proximal; Arthroplasty, Replacement, Shoulder; Reverse Total Shoulder Arthroplasty; Shoulder Hemiarthroplasty
MeSH Terms: conditions — Shoulder Fractures | interventions — Hemiarthroplasty

ARMS (2):
- Reverse Total Shoulder Arthroplasty (Experimental)
  Interventions: Procedure: Reverse Total Shoulder Arthroplasty
- Hemiarthroplasty (Active Comparator)
  Interventions: Procedure: Hemiarthroplasty

INTERVENTIONS:
Procedure: Reverse Total Shoulder Arthroplasty
  Arms: Reverse Total Shoulder Arthroplasty
Procedure: Hemiarthroplasty
  Arms: Hemiarthroplasty

SUMMARY:
Proximal humeral fractures are common injuries with the highest incidence being amongst the elderly. Most proximal humeral fractures are nondisplaced or minimally displaced. The majority of these are reliably treated nonoperatively with an acceptable functional outcome. The treatment of displaced fractures is more controversial. Consensus is lacking as to when surgery is indicated or what type of procedure to choose if surgery is elected. Displaced 3- and 4-part fractures where internal fixation is deemed unreliable have been considered an indication for hemiarthroplasty. Hemiarthroplasty gives reasonable control of pain but the resulting shoulder function and range of motion is unpredictable. The use of reverse total shoulder arthroplasty is increasing and might result in a better range of motion then hemiarthroplasty.

The aim of this multicenter study is to test the hypothesis that reverse total shoulder arthroplasty gives better shoulder function than hemiarthroplasty for displaced 3- and 4-part proximal humeral fractures.

ELIGIBILITY:
Inclusion criteria

* Displaced 3- or 4-part fracture of the proximal humerus
* Age over 70 years
* Independent living
* Low energy trauma

Exclusion criteria

* Pre-existing shoulder disease
* Severe cognitive dysfunction
* More than 14 days from injury to surgery
* Comorbidity that affects shoulder rehabilitation considerably
* Concurrent injury that affect shoulder rehabilitation considerably

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Dates: Start 2013-09-10 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2020-09-02 (Actual)

PRIMARY OUTCOMES:
Constant-Murley Score | 24 months
  The Constant-Murley score is used to assess shoulder function. The maximum score is 100 points. Higher scores represent better shoulder function.
WOOS (Western Ontario Osteoarthritis of the Shoulder) Index | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Per Olerud, MD, Principal Investigator — Karolinska Institutet; Carl Ekholm, MD, Study Director — Sahlgrenska Academy

REFERENCES:
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196